CLINICAL TRIAL: NCT00477490
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Group, Multi-Center Study With a Double Blind Extension Investigating the Efficacy and Safety of a Fast- Dissolving ("Melt") Formulation of Desmopressin for the Treatment of Nocturia in Adults
Brief Title: Efficacy and Safety of Desmopressin Melt for the Treatment of Nocturia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FE992026 CS29
Record Dates: First submitted 2007-05-22; First posted 2007-05-23 (Estimated); Results first posted 2015-11-02 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-09

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): Participants took a placebo 'melt' for 28 days to complete part 1 of the study. In part 2, placebo patients were randomized to one of the other 4 treatment arms based on assignments predetermined at the initial randomization, to receive active desmopressin melt for between 1 and 6 months (until the database for part 1 was locked and treatment was unblinded).
  Interventions: Drug: Placebo
- desmopressin melt 10 μg (Experimental): Participants took desmopressin melt 10 μg for 28 days to complete part 1 of the study. Participants continued on this dose in part 2 of the study for between 1 and 6 months (until the database for part 1 was locked and treatment was unblinded).
  Interventions: Drug: desmopressin acetate
- desmopressin melt 25 μg (Experimental): Participants took desmopressin melt 25 μg for 28 days to complete part 1 of the study. Participants continued on this dose in part 2 of the study for between 1 and 6 months (until the database for part 1 was locked and treatment was unblinded).
  Interventions: Drug: desmopressin acetate
- desmopressin melt 50 μg (Experimental): Participants took desmopressin melt 50 μg for 28 days to complete part 1 of the study. Participants continued on this dose in part 2 of the study for between 1 and 6 months (until the database for part 1 was locked and treatment was unblinded).
  Interventions: Drug: desmopressin acetate
- desmopressin melt 100 μg (Experimental): Participants will take desmopressin melt 100 μg for 28 days to complete part 1 of the study. Participants will continue on this dose in part 2 of the study for between 1-6 months (until the database for part 1 is locked and treatment is unblinded).
  Interventions: Drug: desmopressin acetate

INTERVENTIONS:
Drug: desmopressin acetate — Oral lyophilisate of desmopressin acetate placed under the participant's tongue, without water, once daily approximately 1 hour before bedtime in the assigned dosage: 10, 25, 50 or 100 μg
  Other Names: Minirin® Melt; Nocturin®; FE992026
  Arms: desmopressin melt 10 μg; desmopressin melt 100 μg; desmopressin melt 25 μg; desmopressin melt 50 μg
Drug: Placebo — Oral placebo placed under the participant's tongue, without water, once daily approximately 1 hour before bedtime.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of several doses of the melt formulation of desmopressin in a broad population of adult patients with nocturia.

ELIGIBILITY:
Inclusion Criteria

1. Written informed consent prior to the performance of any study-related activity.
2. Patients 18 years and older with an average of ≥ 2 nocturnal voids per night as determined by a 3 day frequency-volume chart during the screening period.

Exclusion Criteria:

Males:

1. Clinical suspicion of bladder outlet obstruction and/or urine flow < 5 ml/s. If medical history and/or physical examination suggest bladder outlet obstruction, uroflowmetry should be performed to confirm the diagnosis
2. Surgical treatment for bladder outlet obstruction/benign prostatic hyperplasia performed within the past 6 months

   Females:
3. Pregnancy. Females of reproductive age must have documentation of a reliable method of contraception.
4. Use of pessary for pelvic prolapse.
5. Unexplained pelvic mass.

   Males and Females:
6. Clinical suspicion of urinary retention and/or post void residual volume > 150 ml. If medical history and/or physical examination suggest urinary retention, bladder ultrasound or catheterization should be performed to confirm the diagnosis.
7. Current or past urologic malignancy (e.g., bladder cancer, prostate cancer).
8. Clinical evidence of current genitourinary tract pathology that could interfere with voiding.
9. History of neurogenic detrusor activity (previously known as detrusor hyperreflexia).
10. Suspicion or evidence of cardiac failure.
11. Uncontrolled hypertension.
12. Uncontrolled diabetes mellitus.
13. Renal insufficiency. Serum creatinine must be within normal limits and estimated glomerular filtration rate (eGFR) >=60 mL/min.
14. Active hepatic and/or biliary disease. Aspartate transaminase (AST) or alanine transaminase (ALT) should not be >2 times the upper limit of normal. Total bilirubin should not be > 1.5 mg/dL.
15. Hyponatremia. Serum sodium level must be within normal limits
16. Syndrome of Inappropriate antidiuretic hormone secretion (SIADH).
17. Diabetes insipidus (urine output > 40 ml/kg over 24 hours) as determined by the 3-day voiding diary.
18. Psychogenic or habitual polydipsia
19. Obstructive sleep apnea

    Other
20. Known alcohol or substance abuse
21. Work or lifestyle potentially interfering with regular nighttime sleep (e.g., shift workers)
22. Previous desmopressin treatment for nocturia.
23. Any other medical condition, laboratory abnormality, psychiatric condition, mental incapacity or language barrier that, in the judgment of the investigator, could impair patient participation in the trial.
24. Use of loop diuretics (furosemide, torsemide, ethacrynic acid). Other classes of diuretics (thiazides, triamterene, chlorthalidone, amiloride, indapamide) were permitted, either as monotherapy or combination therapy. Subjects using a diuretic were to be encouraged to take it in the morning, if medically feasible.
25. Use of any other investigational drug within 30 days of screening.

Concomitant Medications

The following medications are permitted provided that the subject has been on a stable dose for the 3 months prior to the screening date (i.e. treatment has not been initiated or discontinued and there has been no change in dose):

* Alpha-blockers: Cardura (doxazosin); Flomax (tamsulosin); Hytrin (terazosin); Uroxatral (alfuzosin)
* 5 alpha-reductase inhibitors: Avodart (dutasteride); Proscar (finasteride)
* Antispasmodic, anticholinergic, antimuscarinic therapy for overactive bladder: Detrol, Detrol LA (tolterodine); Ditropan, Ditropan XL (oxybutynin); Enablex (darifenacin); Levsin(hyoscyamine); Oxytrol transdermal (oxybutynin); Sanctura (trospium); Vesicare (solifenacin)
* Sedative/hypnotic medications for sleep disorders
* Selective serotonin and mixed norepinephrine/serotonin reuptake inhibitors: Celexa (citalopram); Cymbalta (duloxetine); Effexor (venlafaxine); Lexapro (escitalopram); Paxil(paroxetine); Prozac (fluoxetine); Zoloft (sertraline)
* Chronic use of nonsteroidal anti-inflammatory agents
* Diabinese (chlorpropamide)
* Carbamazepine (carbatrol/tegretol)
* Amiodarone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 799 (Actual)
Dates: Start 2007-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (80):
- United States (70):
  - Radiant Research, Birmingham, Alabama
  - Radiant Research, Scottsdale, Arizona
  - Arkansas Primary Care Clinic, Little Rock, Arkansas
  - Advanced Urology Medical Center, Anaheim, California
  - Impact Clinical Trials, Beverly Hills, California
  - Atlantic Urology Medical Group, Long Beach, California
  - California Professional Research, Newport Beach, California
  - San Diego Uro-Research, San Diego, California
  - Radiant Research, Santa Rosa, California
  - West Coast Clinical Research, Tarzana, California
  - Western Clinical Research, Torrance, California
  - Urology Associates PC, Denver, Colorado
  - Downtown Women's Health Care, Denver, Colorado
  - Genitourinary Surgical Consultants, Denver, Colorado
  - Connecticut Clinical Research Center, LLC, Middlebury, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - Medsearch Professional Group, Miami, Florida
  - Sunrise Medical Research, Plantation, Florida
  - Radiant Research, Stuart, Florida
  - Southeastern Research Group, Inc., Tallahassee, Florida
  - Tampa Bay Urology, Tampa, Florida
  - Radiant Research, West Palm Beach, Florida
  - Southeastern Medical Research Institute, Columbus, Georgia
  - Investigational site - PC, Dunwoody, Georgia
  - Accelovance, Peoria, Illinois
  - Radiant Research, Kansas City, Overland Park, Kansas
  - Benchmark Research, Metairie, Louisiana
  - Regional Urology, LLC, Shreveport, Louisiana
  - Pierremont Women's Clinic, Shreveport, Louisiana
  - FutureCare Studies, Inc., Springfield, Massachusetts
  - Radiant Research Inc., St Louis, Missouri
  - Women's Clinic of Lincoln, P.C, Lincoln, Nebraska
  - Investigational site, Las Vegas, Nevada
  - AdvanceMed Research, Lawrenceville, New Jersey
  - Lawrenceville Urology, Lawrenceville, New Jersey
  - Morristown Urology, Morristown, New Jersey
  - Urology Group of New Mexico, PC, Albuquerque, New Mexico
  - Upstate Urology, Albany, New York
  - Investigational site - Adult & Pediatric Urology, Carmel, New York
  - AccuMed Research Associates, Garden City, New York
  - University Urology Associates, New York, New York
  - Ferring Pharmaceutical Inc, Suffern, New York
  - Northeast Urology Research, Concord, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - New Hanover Medical Research, Wilmington, North Carolina
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Radiant Research, Cincinnati, Ohio
  - Radiant Research - Akron, Mogadore, Ohio
  - Urologic Consultants of SE PA, Bala-Cynwyd, Pennsylvania
  - Philadelphia Clinical Research, LLC, Philadelphia, Pennsylvania
  - Radiant Research, Philadelphia, Pennsylvania
  - Advanced Clinical Concepts, Reading, Pennsylvania
  - University Medical Group, Greenville, South Carolina
  - Radiant Research, Greer, Greer, South Carolina
  - Palmetto Medical Research, Mt. Pleasant, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Holston Medical Group, Kingsport, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Advanced Research Associates, Corpus Christi, Texas
  - Health Central Women's Care, Dallas, Texas
  - Accelovance, Houston, Texas
  - Regional Medical Center and Diagnostic, Humble, Texas
  - Radiant Research San Antonio, San Antonio, Texas
  - Urology San Antonio Research, PA, San Antonio, Texas
  - Virginia Urology Center, Richmond, Virginia
  - Urology of Virginia PC, Virginia Beach, Virginia
  - Women's Clinical Research Center, Seattle, Washington
  - Investigational site - Medical Professional, Seattle, Washington
  - Seattle Urology Research Center, Seattle, Washington
- Canada (10):
  - Southern Interior Medical Center, Kelowna, British Columbia
  - Can-Med Clinical Research Inc., Victoria, British Columbia
  - Investigational site - Clinical Research, Victoria, British Columbia
  - Investigational site - Professional Corporation, Fredericton, New Brunswick
  - The Male/Female Health and Reserach, Barrie, Ontario
  - Brantford Urology Research, Brantford, Ontario
  - Guelph Urology Associates, Guelph, Ontario
  - Investigational site, North Bay, Ontario
  - The Fe/Male Health Centres, Oakville, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

REFERENCES:
- [Background] Juul KV, Klein BM, Norgaard JP. Long-term durability of the response to desmopressin in female and male nocturia patients. Neurourol Urodyn. 2013 Apr;32(4):363-70. doi: 10.1002/nau.22306. Epub 2012 Sep 12. PMID 22972524
- [Result] Weiss JP, Zinner NR, Klein BM, Norgaard JP. Desmopressin orally disintegrating tablet effectively reduces nocturia: results of a randomized, double-blind, placebo-controlled trial. Neurourol Urodyn. 2012 Apr;31(4):441-7. doi: 10.1002/nau.22243. Epub 2012 Mar 22. PMID 22447415
- [Derived] Juul KV, Malmberg A, van der Meulen E, Walle JV, Norgaard JP. Low-dose desmopressin combined with serum sodium monitoring can prevent clinically significant hyponatraemia in patients treated for nocturia. BJU Int. 2017 May;119(5):776-784. doi: 10.1111/bju.13718. Epub 2016 Dec 10. PMID 27862898
- [Derived] Bliwise DL, Holm-Larsen T, Goble S. Increases in duration of first uninterrupted sleep period are associated with improvements in PSQI-measured sleep quality. Sleep Med. 2014 Oct;15(10):1276-8. doi: 10.1016/j.sleep.2014.05.013. Epub 2014 Jun 13. PMID 25172115
- [Derived] Juul KV, Klein BM, Sandstrom R, Erichsen L, Norgaard JP. Gender difference in antidiuretic response to desmopressin. Am J Physiol Renal Physiol. 2011 May;300(5):F1116-22. doi: 10.1152/ajprenal.00741.2010. Epub 2011 Mar 2. PMID 21367921

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighty-eight (88) sites were initiated in the United States and Canada, and 81 of these sites screened subjects; 78 sites enrolled and randomized subjects.
  A total of 1412 subjects were screened for Part I of the study; 613 subjects were screening failures.
Pre-assignment Details: Potential subjects were given a sleep/voiding diary and urine collection device to record the time and volume of each void for 3 consecutive 24-hour periods.
  Randomization was stratified by age (<65, ≥65 years) and by the absence/presence of nocturnal polyuria, defined as a ratio of nighttime urine volume/24-hour urine volume ≥33%.
Groups:
- Placebo: Participants took a placebo 'melt' for 28 days to complete Part I of the study. In Part II, placebo patients were randomized to one of the other four treatment arms to receive active desmopressin melt for between 1-6 months (until the database for Part I was locked and treatment was unblinded).
- Desmopressin Melt 10 μg: Participants took desmopressin melt 10 μg for 28 days to complete Part I of the study. Participants continued this dose in study Part II for between 1-6 months (until the database for Part I was locked and treatment was unblinded).
- Desmopressin Melt 25 μg: Participants took desmopressin melt 25 μg for 28 days to complete Part I of the study. Participants continued this dose in study Part II for between 1-6 months (until the database for Part I was locked and treatment was unblinded).
- Desmopressin Melt 50 μg: Participants took desmopressin melt 50 μg for 28 days to complete Part I of the study. Participants continued this dose in study Part II for between 1-6 months (until the database for Part I was locked and treatment was unblinded).
- Desmopressin Melt 100 μg: Participants took desmopressin melt 100 μg for 28 days to complete Part I of the study. Participants continued this dose in study Part II for between 1-6 months (until the database for Part I was locked and treatment was unblinded).
- Placebo to 10 μg: Participants randomized to Placebo in study Part I were re-randomized to receive active desmopressin in Part II. These participants were randomized to receive desmopressin melt 10 μg once daily about an hour before bedtime.
- Placebo to 25 μg: Participants randomized to Placebo in study Part I were re-randomized to receive active desmopressin in Part II. These participants were randomized to receive desmopressin melt 25 μg once daily about an hour before bedtime.
- Placebo to 50 μg: Participants randomized to Placebo in study Part I were re-randomized to receive active desmopressin in Part II. These participants were randomized to receive desmopressin melt 50 μg once daily about an hour before bedtime.
- Placebo to 100 μg: Participants randomized to Placebo in study Part I were re-randomized to receive active desmopressin in Part II. These participants were randomized to receive desmopressin melt 100 μg once daily about an hour before bedtime.
Period: Part I: 4 Week Efficacy
Arm/Group | Placebo | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg | Placebo to 10 μg | Placebo to 25 μg | Placebo to 50 μg | Placebo to 100 μg
Started | 160 | 163 | 158 | 158 | 160 | 0 | 0 | 0 | 0
ITT Population | 156 (Received at least one dose of study drug and provided at least one primary efficacy measure.) | 155 (Received at least one dose of study drug and provided at least one primary efficacy measure.) | 152 (Received at least one dose of study drug and provided at least one primary efficacy measure.) | 148 (Received at least one dose of study drug and provided at least one primary efficacy measure.) | 146 (Received at least one dose of study drug and provided at least one primary efficacy measure.) | 0 | 0 | 0 | 0
Completed | 145 | 144 | 148 | 138 | 135 | 0 | 0 | 0 | 0
Not Completed | 15 | 19 | 10 | 20 | 25 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 4 | 0 | 5 | 6 | 0 | 0 | 0 | 0
Not completed — Serum Sodium <= 125mmol/L | 1 | 0 | 0 | 5 | 4 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 5 | 6 | 4 | 9 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 4 | 1 | 5 | 3 | 0 | 0 | 0 | 0
Not completed — Other, not specified | 2 | 4 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Not Reported | 1 | 2 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Period: Part II: Extension Week 5 up to Day 169
Arm/Group | Placebo | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg | Placebo to 10 μg | Placebo to 25 μg | Placebo to 50 μg | Placebo to 100 μg
Started | 0 | 135 | 135 | 132 | 127 | 31 | 37 | 34 | 34
Completed | 0 | 107 | 120 | 120 | 107 | 25 | 32 | 29 | 26
Not Completed | 0 | 28 | 15 | 12 | 20 | 6 | 5 | 5 | 8
Not completed — Withdrawal by Subject | 0 | 15 | 7 | 7 | 10 | 4 | 2 | 3 | 2
Not completed — Adverse Event | 0 | 2 | 3 | 1 | 1 | 1 | 1 | 1 | 4
Not completed — Lost to Follow-up | 0 | 3 | 2 | 0 | 5 | 0 | 1 | 0 | 0
Not completed — Decreased sodium | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Excluded medication | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other, not specified | 0 | 4 | 2 | 4 | 2 | 1 | 1 | 0 | 1
Not completed — Not reported | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Demographic data offered from the Intent-to-Treat population
Groups:
- Placebo: Participants took a placebo 'melt' for 28 days to complete Part I of the study. In Part II, placebo patients were randomized to one of the other four treatment arms to receive active desmopressin melt for between 1-6 months (until the database for part 1 was locked and treatment was unblinded).
- Desmopressin Melt 10 μg: Participants took desmopressin melt 10 μg for 28 days to complete Part I of the study. Participants continued on this dose in study Part II for between 1-6 months (until the database for Part I was locked and treatment was unblinded).
- Desmopressin Melt 25 μg: Participants took desmopressin melt 25 μg for 28 days to complete Part I of the study. Participants continued on this dose in study Part II for between 1-6 months (until the database for Part I was locked and treatment was unblinded).
- Desmopressin Melt 50 μg: Participants took desmopressin melt 50 μg for 28 days to complete Part I of the study. Participants continued on this dose in study Part II for between 1-6 months (until the database for Part I was locked and treatment was unblinded).
- Desmopressin Melt 100 μg: Participants took desmopressin melt 100 μg for 28 days to complete Part I of the study. Participants continued on this dose in study Part II for between 1-6 months (until the database for Part I was locked and treatment was unblinded).
- Total: Total of all reporting groups
Arm/Group | Placebo | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg | Total
Number analyzed (Participants) | 156 | 155 | 152 | 148 | 146 | 757
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (13.39) | 61.7 (14.41) | 62.4 (13.22) | 61.6 (11.80) | 62.1 (12.34) | 62.0 (13.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 73 | 65 | 71 | 66 | 341
  Male | 90 | 82 | 87 | 77 | 80 | 416
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 136 | 123 | 120 | 119 | 111 | 609
  Black/African American | 16 | 21 | 28 | 24 | 27 | 116
  Asian | 3 | 2 | 2 | 3 | 6 | 16
  American Indian/Alaskan Native | 0 | 2 | 0 | 0 | 0 | 2
  Native Hawaiian/other Pacific Islander | 0 | 1 | 1 | 0 | 0 | 2
  Other | 1 | 6 | 1 | 2 | 2 | 12
Ethnic Origin [Number; unit: participants]
  Hispanic | 13 | 10 | 10 | 13 | 6 | 52
  Not Hispanic | 143 | 145 | 142 | 135 | 140 | 705

OUTCOME MEASURES:

1. Primary Outcome: Part I: Change From Baseline in Mean Number of Nocturnal Voids at Week 4
Description: The number of nocturnal voids was the average over 3 consecutive 24-hours periods prior to Day 1 and prior to the week 4 visit as recorded in participant diaries.
  This was the first co-primary outcome.
Time Frame: - Week 3 to Day 1 (Baseline), Week 4 (end of Part I)
Population: Intent to treat (ITT) population --All randomized participants who received at least one dose of study drug and provided at least one primary efficacy measure (i.e., nocturnal voids) during Part I were included in the ITT analysis dataset
Measure: Mean (Standard Deviation); unit: nocturnal voids
Arm/Group | Placebo | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg
Number analyzed (Participants) | 156 | 155 | 152 | 148 | 146
nocturnal voids | -0.86 (1.054) | -0.83 (1.069) | -1.00 (1.125) | -1.18 (1.187) | -1.43 (1.219)
Statistical Analysis 1: Comparison: Placebo vs Desmopressin Melt 10 μg; Test type: Superiority or Other; p = 0.9303, ANCOVA — The a priori statistically significant difference versus placebo is p≤0.05; Treatment difference and 95% CI were adjusted for age, absence/presence of nocturnal polyuria, and baseline number of nocturnal voids; Mean Difference (Final Values) = 0.010, 95% CI 2-sided [-0.221 to 0.242]
Statistical Analysis 2: Comparison: Placebo vs Desmopressin Melt 25 μg; Test type: Superiority or Other; p = 0.3104, ANCOVA — The a priori statistically significant difference versus placebo is p≤0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.120, 95% CI 2-sided [-0.353 to 0.112]
Statistical Analysis 3: Comparison: Placebo vs Desmopressin Melt 50 μg; The trial was to be declared positive only if in the 100 μg group, a statistically significant positive effect as compared to placebo on both co-primaries was demonstrated. And only then, the next higher dose group (i.e., 50 μg) could be claimed superior to placebo, if it showed a statistically significant improvement over placebo on both co-primaries; Test type: Superiority or Other; p = 0.0207, ANCOVA — The a priori statistically significant difference versus placebo is p≤0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.277, 95% CI 2-sided [-0.511 to -0.042]
Statistical Analysis 4: Comparison: Placebo vs Desmopressin Melt 100 μg; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p < 0.0001, ANCOVA — The a priori statistically significant difference versus placebo is p≤0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.613, 95% CI 2-sided [-0.848 to -0.378]

2. Primary Outcome: Part I: Percentage of Participants With Greater Than 33 Percent Reduction From Baseline in Mean Number of Nocturnal Voids at Week 4
Description: Percentage of participants in each treatment arm that had a greater than 33% reduction from baseline to the end of Part I (week 4) in mean number of nocturnal voids. Nocturnal void data were recorded in participant diaries.
  This was the second co-primary outcome.
Time Frame: - Week 3 to Day 1 (Baseline), Week 4 (end of Part I)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg
Number analyzed (Participants) | 156 | 155 | 152 | 148 | 146
percentage of participants | 47 | 47 | 50 | 53 | 71
Statistical Analysis 1: Comparison: Placebo vs Desmopressin Melt 10 μg; Test type: Superiority or Other; p = 0.9420, Regression, Logistic — The a priori statistically significant difference versus placebo is p≤0.05; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.017, 95% CI 2-sided [0.647 to 1.598]
Statistical Analysis 2: Comparison: Placebo vs Desmopressin Melt 25 μg; Test type: Superiority or Other; p = 0.5527, Regression, Logistic — The a priori statistically significant difference versus placebo is p≤0.05; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.147, 95% CI 2-sided [0.729 to 1.807]
Statistical Analysis 3: Comparison: Placebo vs Desmopressin Melt 50 μg; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.2662, Regression, Logistic — The a priori statistically significant difference versus placebo is p≤0.05; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.296, 95% CI 2-sided [0.821 to 2.050]
Statistical Analysis 4: Comparison: Placebo vs Desmopressin Melt 100 μg; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — The a priori statistically significant difference versus placebo is p≤0.05; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.893, 95% CI 2-sided [1.795 to 4.715]

3. Secondary Outcome: Part II: Change From Baseline in Mean Number of Nocturnal Voids to Days 29, 57, 113 and 169
Description: Part II outcomes tested the durability of the effect observed in Part I. The number of nocturnal voids was the average over 3 consecutive 24-hours periods prior to Part I baseline and prior to the Part II visit as recorded in participant diaries.
Time Frame: - Week 3 to Day 1 (Baseline), Days 29, 57, 113 and 169
Population: Observed Cases (OC) Analysis Set which consisted of participants who had information on mean number of nocturnal voids for both the screening visit and the final visit in Part I (Day 28) and did not have any major protocol deviations.
Measure: Mean (Standard Deviation); unit: nocturnal voids
Arm/Group | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg | Placebo to 10 μg | Placebo to 25 μg | Placebo to 50 μg | Placebo to 100 μg
Number analyzed (Participants) | 104 | 100 | 93 | 104 | 22 | 28 | 27 | 22
nocturnal voids
  Day 29 (n=104,100,93,104,22,28,27,22) | -1.12 (1.161) | -1.31 (1.163) | -1.43 (1.273) | -1.47 (1.080) | -1.20 (0.912) | -1.19 (1.215) | -1.00 (1.140) | -1.58 (1.169)
  Day 57 (n=86,85,78,81,17,24,21,16) | -1.14 (1.147) | -1.42 (1.231) | -1.50 (1.156) | -1.74 (1.036) | -1.08 (0.618) | -1.53 (1.183) | -1.03 (1.264) | -1.35 (1.363)
  Day 113 (n=53,56,49,47,11,15,13,11) | -1.31 (1.195) | -1.56 (1.158) | -1.65 (1,279) | -1.95 (1.088) | -0.76 (0.870) | -1.67 (1.039) | -1.21 (1.085) | -1.76 (1.193)
  Day 169 (n=17,15,17,15,3,3,4,2) | -1.47 (1.537) | -1.71 (1.214) | -1.65 (0.916) | -1.76 (0.801) | -1.78 (0.192) | -2.00 (2.000) | -2.33 (0.272) | -2.50 (1.179)

4. Secondary Outcome: Part II: Percentage of Participants With Greater Than 33 Percent Reduction From Baseline in Mean Number of Nocturnal Voids to Days 29, 57, 113 and 169
Description: Part II outcomes tested the durability of the effect observed in Part I. Percentage of participants in each treatment arm that had a greater than 33% reduction from baseline to Days 29, 57, 113 and 169 in mean number of nocturnal voids. Nocturnal void data were recorded in participant diaries.
Time Frame: - Week 3 to Day 1 (Baseline), Days 29, 57, 113 and 169
Population: Observed Cases (OC) Analysis Set which consisted of participants who had information on mean number of nocturnal voids for both the screening visit and the final visit in Part I (Day 28) and did not have any major protocol deviations. Participants had data representing the visit.
Measure: Number; unit: percentage of participants
Arm/Group | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg | Placebo to 10 μg | Placebo to 25 μg | Placebo to 50 μg | Placebo to 100 μg
Number analyzed (Participants) | 104 | 100 | 93 | 104 | 22 | 28 | 27 | 22
percentage of participants
  Day 29 (n=104,100,93,104,22,28,27,22) | 57 | 64 | 68 | 68 | 73 | 43 | 48 | 73
  Day 57 (n=86,85,78,81,17,24,21,16) | 59 | 68 | 71 | 83 | 41 | 71 | 43 | 69
  Day 113 (n=53,56,49,47,11,15,13,11) | 58 | 79 | 69 | 87 | 55 | 73 | 54 | 73
  Day 169 (n=17,15,17,15,3,3,4,2) | 61 | 80 | 76 | 87 | 100 | 67 | 100 | 100

5. Secondary Outcome: Part I: Change From Baseline in Total Reported Sleep Time at Week 4
Description: Total sleep time was recorded by participants in study diaries.
Time Frame: - Week 3 to Day 1 (Baseline), Week 4 (end of Part I)
Population: Intent to treat (ITT) population --All randomized subjects who received at least one dose of study drug and provided at least one primary efficacy measure (i.e., number of nocturnal voids) during Part I were included in the ITT analysis dataset. Participants analyzed had baseline and Week 4/Day 28/End of Part 1 measurements.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg
Number analyzed (Participants) | 139 | 137 | 141 | 138 | 133
minutes | 24.6 (80.66) | 7.8 (58.55) | 15.9 (53.92) | 24.9 (72.21) | 19.0 (68.94)

6. Secondary Outcome: Part I: Change From Baseline in Initial Period of Undisturbed Sleep at Week 4
Description: Initial period of undisturbed sleep was the time elapsed from first falling asleep until either first void or morning arising. Data were captured in patient diaries.
Time Frame: - Week 3 to Day 1 (Baseline), Week 4 (end of Part I)
Population: ITT population --All randomized subjects who received at least one dose of study drug and provided at least one primary efficacy measure (i.e., number of nocturnal voids) during Part I were included in the ITT analysis dataset. Participants with both baseline and Week 4/Day 28/End of Part I data are included.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg
Number analyzed (Participants) | 126 | 126 | 121 | 123 | 121
minutes | 38.7 (88.79) | 50.9 (111.47) | 82.7 (105.57) | 85.1 (109.33) | 106.7 (116.18)

7. Secondary Outcome: Part I: Change From Baseline in Quality of Life Assessed by The International Consultation on Incontinence Modular Questionnaire - Nocturia (ICIQ-N) at Week 4
Description: The ICIQ-N is a self-administered questionnaire designed to assess the frequency and bother of daytime and nighttime urination. Subjects were asked to rate the degree of bother of daytime urination and nighttime urination on a scale ranging from 0 (not at all) to 10 (a great deal). Higher numbers indicate lower quality of life.
Time Frame: - Week 3 to Day 1 (Baseline), Week 4 (end of Part I)
Population: Intent to treat population of participants who completed the questionnaire at both baseline and end of Part 1.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg
Number analyzed (Participants) | 147 | 145 | 143 | 137 | 137
units on a scale
  Daytime urination: How much does it bother you? | -0.7 (2.61) | -0.7 (2.59) | -0.9 (2.96) | -0.7 (2.86) | -1.0 (2.90)
  Nighttime urination: How much does it bother you? | -1.4 (2.86) | -1.8 (2.96) | -2.1 (3.19) | -2.2 (3.33) | -2.5 (3.32)

8. Secondary Outcome: Part I: Change From Baseline in the Two Domain Scores of the Nocturia Quality of Life (NQoL) Questionnaire at Week 4
Description: The NQoL questionnaire is a self-administered questionnaire designed to assess the impact of nocturia on quality of life. It contains a sleep/energy domain (6 questions), a bother/concern domain (6 questions), and 1 global QoL question. The twelve core questions are scored on a 0 to 4 scale with higher numbers indicating a better quality of life. Domain summary scores were calculated by transforming the raw score into a 0-100 scale with higher numbers indicating a better quality of life.
Time Frame: - Week 3 to Day 1 (Baseline), Week 4 (end of Part I)
Population: Intent to treat population of participants who completed the questionnaire at both baseline and end of Part 1.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg
Number analyzed (Participants) | 147 | 148 | 145 | 135 | 138
units on a scale
  Sleep/Energy Domain | 15.2 (19.30) | 12.3 (23.54) | 14.6 (18.71) | 14.7 (20.92) | 16.3 (21.09)
  Bother/Concern Domain | 12.7 (19.73) | 14.7 (23.42) | 15.7 (21.29) | 15.2 (25.46) | 18.2 (23.29)

9. Secondary Outcome: Part I: Change From Baseline in Quality of Sleep as Assessed by the Global Score of the Pittsburgh Sleep Quality Index (PSQI) at Week 4
Description: The PSQI is a self-administered 19-item questionnaire designed to assess sleep quality and disturbances. The global score ranges from 0 (better sleep quality) to 21 (worse sleep quality). Higher numbers indicate lower quality of life.
Time Frame: - Week 3 to Day 1 (Baseline), Week 4 (end of Part I)
Population: Intent to treat population of participants who completed the questionnaire at both baseline and end of Part 1.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg
Number analyzed (Participants) | 143 | 138 | 136 | 129 | 132
units on a scale | -1.6 (2.8) | -1.6 (2.8) | -1.8 (3.0) | -2.0 (3.2) | -1.9 (3.0)

10. Secondary Outcome: Part I: Change From Baseline in the Mental Health Summary and the Physical Health Summary of the Short Form-12 Version 2 (SF-12v2) at Week 4
Description: The SF-12v2 was used to measure the impact of nocturia and lack of sleep on general quality of life. The SF-12 consists of 12 questions. Data were analyzed using norm-based scoring and summarized along 2 dimensions: Physical Health Summary and Mental Health Summary. Each summary has a range from 0 (poor health) to 100 (highest level of health). Higher numbers indicate better quality of life.
Time Frame: - Week 3 to Day 1 (Baseline), Week 4 (end of Part I)
Population: Intent to treat population of participants who completed the questionnaire at both baseline and end of Part 1.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg
Number analyzed (Participants) | 146 | 146 | 140 | 137 | 137
units on a scale
  Mental Health Summary | 2.4 (7.98) | 2.5 (8.06) | 2.1 (8.16) | 2.2 (8.39) | 1.7 (7.73)
  Physical Health Summary | 1.0 (6.81) | 0.5 (6.89) | 1.2 (7.17) | 0.6 (7.10) | 2.3 (6.62)

11. Secondary Outcome: Part I: Participants With Treatment-Emergent Adverse Events (AEs) During Study Part I
Description: A treatment-emergent adverse event (AE) was any AE occurring during the treatment period or a pretreatment AE that worsened in intensity during the treatment period. The treatment period was the period during which a subject received investigational medicinal product. If a subject discontinued the investigational medicinal product, the date of last dose was the last day of the treatment period.
Time Frame: Day 1 up to Week 4 (end of Part I)
Population: Part I Safety Population includes study participants who received study intervention and had at least one safety assessment during study Part I.
Measure: Number; unit: participants
Arm/Group | Placebo | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg
Number analyzed (Participants) | 160 | 163 | 158 | 158 | 160
participants
  All AEs | 94 | 100 | 98 | 103 | 110
  Deaths | 0 | 0 | 0 | 0 | 0
  Serious AEs | 1 | 2 | 1 | 2 | 0
  AEs leading to discontinuation | 8 | 6 | 2 | 13 | 13
  Severe AEs | 4 | 8 | 5 | 13 | 7
  Adverse drug reactions (ADRs) | 62 | 62 | 61 | 73 | 80

12. Secondary Outcome: Part II: Participants With Treatment-Emergent Adverse Events (AEs) During Study Part II
Description: as for outcome 11
Time Frame: Week 5 up to Day 169
Population: Part II Safety Population includes study participants who received study intervention and had at least one safety assessment during study Part II.
Measure: Number; unit: participants
Arm/Group | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg | Placebo to 10 μg | Placebo to 25 μg | Placebo to 50 μg | Placebo to 100 μg
Number analyzed (Participants) | 135 | 135 | 132 | 127 | 31 | 37 | 34 | 34
participants
  All AEs | 95 | 95 | 92 | 100 | 20 | 27 | 25 | 28
  Deaths | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Serious AEs | 3 | 1 | 0 | 2 | 0 | 0 | 2 | 2
  AEs leading to discontinuation | 3 | 3 | 2 | 4 | 1 | 2 | 2 | 5
  Severe AEs | 7 | 4 | 9 | 5 | 1 | 3 | 2 | 1
  Adverse Drug Reactions | 64 | 59 | 58 | 68 | 10 | 16 | 15 | 18

ADVERSE EVENTS:
Time Frame: Part I covers Day 1 to Week 4. Part II covers Week 5 up to Day169.
Groups:
- Part I: Placebo: Participants took a placebo 'melt' for 28 days to complete Part I of the study.
- Part I: Desmopressin Melt 10 μg: Participants took desmopressin melt 10 μg for 28 days to complete Part I of the study.
- Part I: Desmopressin Melt 25 μg: Participants took desmopressin melt 25 μg for 28 days to complete Part I of the study.
- Part I: Desmopressin Melt 50 μg: Participants took desmopressin melt 50 μg for 28 days to complete Part I of the study.
- Part I: Desmopressin Melt 100 μg: Participants took desmopressin melt 100 μg for 28 days to complete Part I of the study. Participants continued on this dose in study Part II for between 1-6 months (until the database for Part I was locked and treatment was unblinded).
- Part II: Desmopressin Melt 10 μg: Participants who took desmopressin melt 10 μg in Part I of the study continued on this dose in Part II which ran between Months 1-6 (until the database for Part I was locked and treatment was unblinded).
- Part II: Desmopressin Melt 25 μg: Participants who took desmopressin melt 25 μg in Part I of the study continued on this dose in Part II which ran between Months 1-6 (until the database for Part I was locked and treatment was unblinded).
- Part II: Desmopressin Melt 50 μg: Participants who took desmopressin melt 50 μg in Part I of the study continued on this dose in Part II which ran between Months 1-6 (until the database for Part I was locked and treatment was unblinded).
- Part II: Desmopressin Melt 100 μg: Participants who took desmopressin melt 100 μg in Part I of the study continued on this dose in Part II which ran between Months 1-6 (until the database for Part I was locked and treatment was unblinded).
- Part II: Placebo to Desmopressin Melt 10 μg: Participants randomized to Placebo in study Part I were re-randomized to receive active desmopressin in Part II. These participants were randomized to receive desmopressin melt 10 μg once daily about an hour before bedtime
- Part II: Placebo to Desmopressin Melt 25 μg: Participants randomized to Placebo in study Part I were re-randomized to receive active desmopressin in Part II. These participants were randomized to receive desmopressin melt 25 μg once daily about an hour before bedtime.
- Part II: Placebo to Desmopressin Melt 50 μg: Participants randomized to Placebo in study Part I were re-randomized to receive active desmopressin in Part II. These participants were randomized to receive desmopressin melt 50 μg once daily about an hour before bedtime.
- Part II: Placebo to Desmopressin Melt 100 μg: Participants randomized to Placebo in study Part I were re-randomized to receive active desmopressin in Part II. These participants were randomized to receive desmopressin melt 100 μg once daily about an hour before bedtime.
Arm/Group | Part I: Placebo | Part I: Desmopressin Melt 10 μg | Part I: Desmopressin Melt 25 μg | Part I: Desmopressin Melt 50 μg | Part I: Desmopressin Melt 100 μg | Part II: Desmopressin Melt 10 μg | Part II: Desmopressin Melt 25 μg | Part II: Desmopressin Melt 50 μg | Part II: Desmopressin Melt 100 μg | Part II: Placebo to Desmopressin Melt 10 μg | Part II: Placebo to Desmopressin Melt 25 μg | Part II: Placebo to Desmopressin Melt 50 μg | Part II: Placebo to Desmopressin Melt 100 μg
Serious Adverse Events (participants affected / at risk) | 1/160 | 2/163 | 1/158 | 2/158 | 0/160 | 3/135 | 1/135 | 0/132 | 2/127 | 0/31 | 0/37 | 2/34 | 2/34
Other Adverse Events (participants affected / at risk) | 64/160 | 67/163 | 62/158 | 76/158 | 79/160 | 71/135 | 69/135 | 66/132 | 73/127 | 17/31 | 23/37 | 19/34 | 20/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part I: Placebo (N=160) | Part I: Desmopressin Melt 10 μg (N=163) | Part I: Desmopressin Melt 25 μg (N=158) | Part I: Desmopressin Melt 50 μg (N=158) | Part I: Desmopressin Melt 100 μg (N=160) | Part II: Desmopressin Melt 10 μg (N=135) | Part II: Desmopressin Melt 25 μg (N=135) | Part II: Desmopressin Melt 50 μg (N=132) | Part II: Desmopressin Melt 100 μg (N=127) | Part II: Placebo to Desmopressin Melt 10 μg (N=31) | Part II: Placebo to Desmopressin Melt 25 μg (N=37) | Part II: Placebo to Desmopressin Melt 50 μg (N=34) | Part II: Placebo to Desmopressin Melt 100 μg (N=34)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adenosquamous cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part I: Placebo (N=160) | Part I: Desmopressin Melt 10 μg (N=163) | Part I: Desmopressin Melt 25 μg (N=158) | Part I: Desmopressin Melt 50 μg (N=158) | Part I: Desmopressin Melt 100 μg (N=160) | Part II: Desmopressin Melt 10 μg (N=135) | Part II: Desmopressin Melt 25 μg (N=135) | Part II: Desmopressin Melt 50 μg (N=132) | Part II: Desmopressin Melt 100 μg (N=127) | Part II: Placebo to Desmopressin Melt 10 μg (N=31) | Part II: Placebo to Desmopressin Melt 25 μg (N=37) | Part II: Placebo to Desmopressin Melt 50 μg (N=34) | Part II: Placebo to Desmopressin Melt 100 μg (N=34)
Dry mouth (Gastrointestinal disorders) | 53 | 53 | 50 | 54 | 49 | 56 | 47 | 46 | 47 | 13 | 14 | 13 | 13
Nausea (Gastrointestinal disorders) | 1 | 4 | 4 | 9 | 10 | 3 | 6 | 5 | 5 | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 5 | 6 | 9 | 3 | 6 | 7 | 10 | 4 | 0 | 2 | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 3 | 2 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 2 | 2 | 2 | 1 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 0 | 1 | 3 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 2 | 0 | 1 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 7 | 4 | 5 | 7 | 1 | 2 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 5 | 4 | 3 | 4 | 1 | 2 | 1 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 3 | 2 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 2
Blood sodium decreased (Investigations) | 1 | 2 | 2 | 4 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 8 | 11 | 2 | 2 | 1 | 7 | 0 | 1 | 2 | 1
Headache (Nervous system disorders) | 11 | 13 | 6 | 15 | 14 | 10 | 11 | 13 | 12 | 1 | 3 | 2 | 2
Dizziness (Nervous system disorders) | 1 | 7 | 3 | 8 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 3 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention